CLINICAL TRIAL: NCT04837495
Title: Stellate Ganglion Block Efficacy in Control of Arrhythmia and Cardiovascular Changes in Addition to, Postoperative Analgesia in Laparoscopic Cholecystectomy
Brief Title: Stellate Ganglion Block in Control of Arrhythmia in Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB17101436
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Arrythmia; Pain, Acute
Keywords: Arrythmia; Acute pain
MeSH Terms: conditions — Arrhythmias, Cardiac; Acute Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stellate Ganglion block group (Active Comparator): will include 20 patients: each one will receive 10 ml lidocaine 2% right stellate ganglion block (RSGB) under sonar guidance
  Interventions: Procedure: right stellate ganglion block
- Control group (No Intervention): will include 20 patients: a control group

INTERVENTIONS:
Procedure: right stellate ganglion block — The skin should be anaesthetised with lidocaine 2%. Using a lateral approach and in-plane imaging, a blunt regional anaesthesia needle should be advanced deep to the carotid sheath towards the longus colli muscle. Following careful aspiration, inject 10 ml lidocaine 2% that will result in expansion of the fascia of the longus colli. Confirmation of the SGB success can be detected by warming of left upper limb and left Horner's syndrome.
  Arms: Stellate Ganglion block group

SUMMARY:
During Laparoscopic cholecystectomy, carbon dioxide (CO2) pneumoperitoneal laparoscopic surgery, CO2-pneumoperitoneum activates the sympathoadrenomedullary system to increase the release of catecholamines such as epinephrine (E) norepinephrine (NE) and dopamine (DA). During stress, E and NE are secreted by the adrenal medulla into blood circulation to promote glycogenolysis to increase blood glucose, speed up lipolysis and accelerate heartbeats. Stellate g anglion block (SGB) reters to the blockade of sympathetic nerves including the large area covered by middle cervical, vertebral arterial. stellate ganglions and ther pre- and post- ganglions. SGB affects both peripheral and central nervous systems. In the peripheral system. the sympathetic pre- and post-ganglionic fibers in the innervated areas of stellate ganglion are affected. Therefore, the control of vascular dilatation and constriction, muscular movement, bronchial smooth muscle relaxation and contraction, and pain conduction, by sympathetic nerves is inhibited. In the central nervous system, the hypothalamus is mainly involved in the regulation of systemic autonomic nervous, immune and endocrine systems, and to maintain homeostasis.

CO2-pneumoperitoneum causes severe stress-related homeostatic disorders including arrhythmia and blood pressure changes. This study will examine the effects of stellate ganglion block (SGB) on hemodynamics and stress response in patients undergoing CO-pneumoperitoneal surgery.

DETAILED DESCRIPTION:
Laparoscopic surgery is being increasingly recognized for its advantages of minimal invasiveness. mild postoperative pain, short length of hospitalization and rapid recovery and is widely used in general surgery, obstetrics. gynecology and urology. Laparoscopic cholecystectomy (LC) has become the gold standard for surgically treating benign diseases of the gallbladder.

During carbon dioxide (CO2) pneumoperitoneal laparoscopic surgery, CO2-pneumoperitoneum activates the sympathoadrenomedullary system to increase the release of catecholamines such as epinephrine (E) norepinephrine (NE) and dopamine (DA). During stress, E and NE are secreted by the adrenal medulla into blood circulation to promote glycogenolysis to increase blood glucose, speed up lipolysis and accelerate heartbeats. Stellate g anglion block (SGB) reters to the blockade of sympathetic nerves including the large area covered by middle cervical, vertebral arterial. stellate ganglions and ther pre- and post- ganglions. SGB affects both peripheral and central nervous systems. In the peripheral system. the sympathetic pre- and post-ganglionic fibers in the innervated areas of stellate ganglion are affected. Therefore, the control of vascular dilatation and constriction, muscular movement, bronchial smooth muscle relaxation and contraction, and pain conduction, by sympathetic nerves is inhibited. In the central nervous system, the hypothalamus is mainly involved in the regulation of systemic autonomic nervous, immune and endocrine systems, and to maintain homeostasis.

CO2-pneumoperitoneum causes severe stress-related homeostatic disorders including arrhythmia and blood pressure changes. This study will examine the effects of stellate ganglion block (SGB) on hemodynamics and stress response in patients undergoing CO-pneumoperitoneal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 -60 years
* american society of anesthesiologists status I-II
* Scheduled for elective laparoscopic cholecystectomy

Exclusion Criteria:

* Patients with chronic renal dysfunction.
* Patients with hypo/hyper-thyroidism.
* Patients with diseases of the autonomic and central nervous systems.
* Patients with cardiopulmonary dysfunction.
* Patients with history of treatment with long-term oral tranquilizers.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Arrhythmia | introperative period
  the incidnese of Arrhythmia

SECONDARY OUTCOMES:
Postoperative pain | 24 hours postoperatively
  Numeric Rating Scale and Visual Analog Scale will be used to evaluate post operative analgesia

CONTACTS AND LOCATIONS:
Locations (1):
- Emad Zarief Kamel Said, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided